CLINICAL TRIAL: NCT01844687
Title: Laboratory Study of the Influence of Oral Cannabidiol on the Subjective, Reinforcing and Cardiovascular Effects of Smoked Marijuana
Brief Title: Laboratory Study of Cannabidiol on the Effects of Smoked Marijuana
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Study Number CBD-001
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2017-04

CONDITIONS: Smoking, Marijuana
Keywords: reinforcement, good drug effect, high, mood, cannabidiol
MeSH Terms: conditions — Marijuana Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Active marijuana (MJ) with 0 mg CBD (Other): Active MJ cigarettes contain 5.30% THC
  Interventions: Drug: CBD
- Active MJ with 200 mg CBD (Other): Active MJ cigarettes contain 5.30% THC
  Interventions: Drug: CBD
- Active MJ with 400 mg CBD (Other): Active MJ cigarettes contain 5.30% THC
  Interventions: Drug: CBD
- Active MJ with 800 mg CBD (Other): Active MJ cigarettes contain 5.30% THC
  Interventions: Drug: CBD
- Inactive MJ with 0 mg CBD (Other): Inactive MJ cigarettes contain 0.01% THC
  Interventions: Drug: CBD
- Inactive MJ with 200 mg CBD (Other): Inactive MJ cigarettes contain 0.01% THC
  Interventions: Drug: CBD
- Inactive MJ with 400 mg CBD (Other): Inactive MJ cigarettes contain 0.01% THC
  Interventions: Drug: CBD
- Inactive MJ with 800 mg CBD (Other): Inactive MJ cigarettes contain 0.01% THC
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — Each subject in the study was tested on eight days, each day receiving a different combination of active/inactive cannabis cigarettes plus 0, 200, 400 or 800 mg of CBD in random order. Cigarettes contained either 0.01 or 5.30% THC. At each visit, participants were given four gelatin capsules containing lactose and 0 or 200 mg of CBD in combinations to achieve scheduled dose level.
  Other Names: cannabidiol is abbreviated CBD

SUMMARY:
The objective of this study is to assess the effects of oral cannabidiol (CBD; 0, 200, 400, 800 mg) on smoked marijuana's (0, 5.6% THC) subjective, reinforcing, cognitive, and cardiovascular effects. This experiment is expected to reveal CBD's intrinsic effects when combined with placebo marijuana, as well as its ability to modulate the behavioral effects of active marijuana.

DETAILED DESCRIPTION:
Marijuana contains many chemicals called cannabinoids. The ingredient mainly responsible for marijuana's psychoactive effects is called THC (delta-9-tetrahydrocannabinol. Another cannabinoid in marijuana is cannabidiol. It is found in smaller quantities than THC. Cannabidiol is thought to interfere with the effects of THC. Therefore, synthetically produced cannabidiol is given to healthy marijuana users in this study to test its capability to reduce the high of THC and, thereby, help to relieve addiction to marijuana.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 50.
* Current marijuana use: Minimum of four times per week, 0.5 joints per occasion during the preceding 4 weeks.
* Able to perform study procedures
* Women practicing an effective form of birth control

Exclusion Criteria:

* Female subjects who are currently pregnant or breastfeeding.
* Current, repeated illicit drug use other than marijuana
* Presence of significant medical illness
* History of heart disease
* Request for drug treatment
* Current parole or probation
* Recent history of significant violent behavior
* Major psychiatric disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, M.D., Principal Investigator — New York State Psychiatric Institute; Robert J Malcolm, M.D., Study Director — Medical University of South Carolina; Sharon Walsh, Ph.D., Study Director — University of Kentucky
Locations (3):
- United States (3):
  - University of Kentucky, Straus Behavioral Research Bldg., 515 Oldham Ct., Lexington, Kentucky
  - Marijuana Outpatient Lab 1051 Riverside Dr. Unit #120, New York, New York
  - Center for Drug and Alcohol Programs, Room 459 North, 67 President St., Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group: Each subject in the study will be tested on eight days, each day receiving a different combination of active/inactive marijuana cigarette plus 0, 200, 400 or 800 mg of cannabidiol
  A subset of study completers will be given 800 mg of cannabidiol on one additional study visit to measure plasma concentrations of cannabidiol for up to 360 minutes after ingestion
Period: Visit 1
Arm/Group | Single Group
Started | 50
Completed | 42
Not Completed | 8
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 5
Period: Visit 2
Arm/Group | Single Group
Started | 42
Completed | 40
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Period: Visit 3
Arm/Group | Single Group
Started | 40
Completed | 35
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — child care problems | 1
Period: Visit 4
Arm/Group | Single Group
Started | 35
Completed | 31
Not Completed | 4
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Period: Visit 5
Arm/Group | Single Group
Started | 31
Completed | 31
Not Completed | 0
Period: Visit 6
Arm/Group | Single Group
Started | 31
Completed | 31
Not Completed | 0
Period: Visit 7
Arm/Group | Single Group
Started | 31
Completed | 31
Not Completed | 0
Period: Visit 8
Arm/Group | Single Group
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: count - only those participants who completed all 8 visits (31)
Arm/Group | Single Group
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 15
  White | 12
  mixed | 4
Region of Enrollment [Number; unit: participants]
  United States | 31
cannabis use (number of days per week) [Mean (Standard Deviation); unit: days per week] | 6.5 (1.0)
cannabis cigarettes per day [Mean (Standard Deviation); unit: cannabis cigarettes used per day] | 5.1 (5.3)
tobacco cigarette smokers [Number; unit: participants] | 18
alcohol drinkers [Number; unit: participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Mood Scale - Subscale 'Feeling High'
Description: Participants rated how much they felt having a "high" feeling from smoked marijuana using a visual analog scale 1-100 mm, 1 (Not at all) - 100 (extremely).
Time Frame: two hours before and after marijuana cigarette smoking
Population: all 31 completers
Measure: Mean (Standard Error); unit: units on a scale VAS 1-100 mm
Groups:
- Active Marijuana (MJ) With 0 mg Cannabidiol (CBD): a placebo comparator measuring the effect of cannabidiol (CBD) on moods produced by smoking 5.30% tetrahydrocannabinol (THC) cannabis cigarettes
- Active MJ With 200 mg CBD: MJ cigarette with 5.3% THC content pretreated with 200 mg CBD
- Active MJ With 400 mg CBD: MJ cigarette with 5.3% THC content pretreated with 400 mg CBD
- Active MJ With 800 mg CBD: MJ cigarette with 5.3% THC content pretreated with 800 mg CBD
- Inactive MJ With 0 mg CBD: MJ cigarette with 0.01% THC content pretreated with 0 mg CBD
- Inactive MJ With 200 mg CBD: MJ cigarette with 0.01% THC content pretreated with 200 mg CBD
- Inactive MJ With 400 mg CBD: MJ cigarette with 0.01% THC content pretreated with 400 mg CBD
- Inactive MJ With 800 mg CBD: MJ cigarette with 0.01% THC content pretreated with 800 mg CBD
Arm/Group | Active Marijuana (MJ) With 0 mg Cannabidiol (CBD) | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
units on a scale VAS 1-100 mm
  -120 mins | 4.35 (2.61) | 2.48 (1.24) | 0.39 (0.18) | 6.55 (2.69) | 0.42 (0.26) | 0.32 (0.19) | 3.35 (2.01) | 1.06 (0.79)
  -30 mins | 4.39 (2.22) | 3.13 (1.75) | 4.32 (1.83) | 2.10 (1.06) | 1.94 (1.37) | 2.00 (1.87) | 1.00 (0.68) | 2.87 (1.87)
  30 mins after MJ | 46.65 (5.69) | 45.90 (5.11) | 43.32 (5.22) | 36.65 (5.37) | 10.52 (2.88) | 17.84 (4.24) | 6.23 (1.56) | 13.94 (3.87)
  60 mins after MJ | 36.55 (5.42) | 38.03 (4.72) | 32.68 (4.79) | 43.10 (5.54) | 7.23 (2.73) | 8.84 (3.08) | 4.03 (1.83) | 6.94 (2.54)
  90 mins after MJ | 24.29 (5.26) | 26.87 (4.28) | 15.39 (3.64) | 24.90 (4.39) | 4.71 (2.25) | 8.39 (2.77) | 2.10 (1.09) | 2.48 (1.27)
  120 mins after MJ | 17.19 (4.60) | 17.13 (3.64) | 11.65 (3.04) | 16.84 (3.89) | 2.35 (1.47) | 4.48 (1.82) | 0.68 (0.33) | 4.26 (2.35)

2. Other Pre Specified Outcome: Marijuana Rating Form - Like
Description: Participants rated how much they liked the effects of smoked marijuana using a visual analog scale 1-100 mm, 1=least, 100= most
Time Frame: 15 - 120 minutes after marijuana cigarette smoking
Population: all study completers
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Active MJ With 0 mg CBD: a placebo comparator measuring the effect of CBD on liking the effects of smoking 5.30% THC cannabis cigarettes
Arm/Group | Active MJ With 0 mg CBD | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
units on a scale
  15 minutes after smoking | 55.32 (5.51) | 65.87 (5.17) | 61.42 (4.92) | 61.94 (5.27) | 25.65 (5.31) | 25.03 (6.05) | 22.81 (5.38) | 22.48 (4.96)
  30 minutes after smoking | 57.10 (5.66) | 57.77 (4.95) | 58.77 (5.84) | 60.58 (5.51) | 20.16 (5.37) | 24.58 (5.71) | 17.97 (4.68) | 18.17 (4.38)
  60 minutes after smoking | 52.55 (6.78) | 57.90 (4.92) | 53.03 (6.08) | 53.26 (6.07) | 14.37 (4.91) | 21.32 (5.65) | 16.03 (5.21) | 23.52 (5.66)
  90 minutes after smoking | 49.58 (6.53) | 51.68 (5.45) | 47.84 (6.50) | 50.13 (5.93) | 15.97 (5.12) | 18.52 (5.57) | 15.06 (4.70) | 17.42 (5.41)
  120 minutes after smoking | 41.29 (6.61) | 46.00 (5.77) | 42.55 (6.62) | 46.81 (6.38) | 14.84 (4.86) | 16.81 (5.21) | 14.00 (5.42) | 16.48 (5.37)

3. Other Pre Specified Outcome: Marijuana Rating Form - Strength
Description: Participants rated the strength effects of smoked marijuana using a visual analog scale 1-100 mm, 1=least, 100= most
Time Frame: 15 - 120 minutes after marijuana cigarette smoking
Population: all study completers
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Active MJ With 0 mg CBD: a placebo comparator measuring the effect of CBD on the strength of effects of smoking 5.30% THC cannabis cigarettes
Arm/Group | Active MJ With 0 mg CBD | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
units on a scale
  15 minutes after smoking | 45.68 (6.19) | 58.03 (4.87) | 51.48 (5.01) | 51.87 (4.99) | 20.32 (4.40) | 20.83 (4.87) | 18.52 (4.52) | 16.87 (3.47)
  30 minutes after smoking | 55.65 (5.30) | 55.03 (4.39) | 48.67 (5.47) | 57.61 (4.75) | 14.42 (3.90) | 18.94 (3.91) | 11.77 (2.80) | 14.83 (3.50)
  60 minutes after smoking | 45.84 (5.77) | 44.68 (4.61) | 39.71 (5.56) | 45.42 (5.18) | 9.03 (3.00) | 13.06 (3.80) | 6.39 (2.58) | 11.65 (3.50)
  90 minutes after smoking | 27.19 (4.92) | 34.97 (5.05) | 28.45 (5.64) | 32.52 (6.11) | 7.03 (2.51) | 11.19 (3.68) | 6.48 (2.81) | 7.94 (3.19)
  120 minutes after smoking | 18.68 (4.39) | 22.87 (4.80) | 19.42 (4.52) | 28.45 (5.81) | 7.55 (3.29) | 8.35 (2.89) | 4.65 (2.59) | 7.19 (3.14)

4. Other Pre Specified Outcome: Optional Additional Puffs of MJ Cigarette
Description: Participants were allowed to choose to take or reject additional puffs of the same type of MJ cigarette they smoked earlier in the day. Counts of participants choosing to take additional puffs are reported.
Time Frame: 150 to 250 minutes after first marijuana cigarette was smoked earlier in the day
Population: all study completers
Measure: Count of Participants; unit: Participants
Groups:
- Active MJ With 0 mg CBD: MJ cigarette with 5.3% THC content pretreated with 0 mg CBD
Arm/Group | Active MJ With 0 mg CBD | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
Participants | 19 | 19 | 18 | 18 | 10 | 11 | 11 | 10

5. Other Pre Specified Outcome: Number of Optional Puffs of MJ Cigarette Taken
Description: Mean number of puffs taken by those participants who chose to take additional puffs.
Time Frame: 150 to 160 minutes after first marijuana cigarette was smoked earlier in the day
Population: Those who took additional puffs of MJ cigarette.
Measure: Mean (Standard Error); unit: number of puffs taken per participant
Arm/Group | Active MJ With 0 mg CBD | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 10 | 11 | 11 | 10
number of puffs taken per participant | 1.68 (0.26) | 1.71 (0.25) | 1.58 (0.26) | 1.55 (0.26) | 0.94 (0.25) | 1.00 (0.25) | 1.00 (0.25) | 0.97 (0.25)

6. Other Pre Specified Outcome: Heart Rate
Description: Heart rate measured at 10 time points, 4 before and 6 after smoking cannabis.
Time Frame: 120 minutes before and 150 minutes after marijuana cigarette smoking
Population: all study completers
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Active MJ With 0 mg CBD | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 31 | 31
beats per minute
  120 minutes before smoking | 66.45 (2.42) | 69.58 (2.39) | 69.90 (2.31) | 66.23 (2.04) | 65.13 (2.09) | 67.65 (1.99) | 65.68 (2.15) | 67.84 (2.19)
  60 minutes before smoking | 68.06 (2.04) | 68.23 (2.22) | 67.87 (2.02) | 67.06 (2.10) | 64.97 (1.78) | 68.32 (1.70) | 65.55 (1.98) | 66.06 (2.09)
  30 minutes before smoking | 65.77 (1.92) | 66.84 (2.37) | 65.42 (1.75) | 66.35 (1.72) | 64.90 (1.62) | 67.42 (1.78) | 67.55 (1.77) | 66.74 (2.22)
  5 minutes before smoking | 60.94 (1.79) | 64.48 (1.97) | 64.55 (1.82) | 65.06 (2.12) | 62.55 (1.67) | 65.58 (1.74) | 63.10 (1.80) | 65.00 (1.98)
  15 minutes after smoking | 78.97 (2.62) | 79.23 (2.44) | 80.74 (2.89) | 78.68 (2.79) | 63.81 (2.03) | 64.16 (1.87) | 63.97 (2.05) | 64.55 (1.79)
  30 minutes after smoking | 71.87 (2.42) | 75.45 (2.36) | 73.03 (2.38) | 75.90 (2.89) | 61.35 (1.77) | 62.94 (1.86) | 62.52 (1.83) | 64.13 (1.72)
  60 minutes after smoking | 64.03 (1.96) | 68.42 (2.60) | 67.94 (2.15) | 68.48 (2.24) | 60.03 (1.72) | 62.03 (1.77) | 61.29 (1.65) | 63.06 (1.89)
  90 minutes after smoking | 65.00 (1.99) | 69.13 (2.19) | 66.16 (2.10) | 68.87 (2.01) | 64.06 (1.80) | 63.97 (1.94) | 61.87 (2.06) | 65.81 (1.94)
  120 minutes after smoking | 69.77 (2.22) | 73.03 (2.30) | 72.90 (2.36) | 70.29 (2.06) | 67.35 (1.90) | 69.68 (2.26) | 67.35 (2.24) | 68.87 (2.14)
  150 minutes after smoking | 67.45 (1.96) | 71.39 (2.18) | 71.03 (2.16) | 68.68 (1.81) | 66.58 (1.69) | 67.71 (1.87) | 66.50 (2.30) | 68.70 (2.11)

7. Other Pre Specified Outcome: Plasma Concentration of CBD
Description: Plasma concentrations of cannabidiol were measured at six time points after oral administration of four 200 mg capsules of CBD.
Time Frame: 6 hours
Population: 8 participants volunteered to come to a ninth session for dosing with 800 mg CBD and donation of 7 blood samples.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Plasma CBD Concentrations: Eight of the 31 participants who completed the study came to a ninth session to receive 800 mg CBD and donate seven blood samples over six hours, one immediately before swallowing CBD capsules, and 6 throughout the next six hours. Plasma samples were analyzed through NIDA contract #NO1DA-14-7788 to David Moody, Ph.D.
Arm/Group | Plasma CBD Concentrations
Number analyzed (Participants) | 8
ng/mL
  baseline | 0 (0)
  60 minutes after dosing | 11.06 (5.43)
  120 minutes after dosing | 38.88 (11.84)
  180 minutes after dosing | 77.95 (25.00)
  240 minutes after dosing | 77.90 (32.72)
  300 minutes after dosing | 50.45 (14.76)
  360 minutes after dosing | 64.04 (23.01)

ADVERSE EVENTS:
Time Frame: Adverse events reported within 72 hours of each cannabidiol administration
Description: Cannabis strength was collapsed for each cannabidiol dose level
Groups:
- Active MJ With 0 mg CBD: 31 subjects were tested with 0 mg CBD and an active marijuana cigarette.
- Active MJ With 200 mg CBD: 31 subjects were tested with 200 mg CBD and an active marijuana cigarette.
- Active MJ With 400 mg CBD: 31 subjects were tested with 400 mg CBD and an active marijuana cigarette.
- Active MJ With 800 mg CBD: 31 subjects were tested with 800 mg CBD and an active MJ cigarette.
- Inactive MJ With 0 mg CBD; Inactive MJ With 200 mg CBD: 31 subjects were tested with 0 mg CBD and an inactive MJ cigarette.
- Inactive MJ With 400 mg CBD: 31 subjects were tested with 400 mg CBD and an inactive marijuana cigarette.
- Inactive MJ With 800 mg CBD: 31 subjects were tested with 800 mg CBD and Inactive MJ cigarette.
  8 of the 31 study completers were given 800 mg of cannabidiol on one additional study visit to measure plasma concentrations of cannabidiol for up to 360 minutes after ingestion. No MJ cigarette was smoked during this session. Adverse events reported during this session are included here.
Arm/Group | Active MJ With 0 mg CBD | Active MJ With 200 mg CBD | Active MJ With 400 mg CBD | Active MJ With 800 mg CBD | Inactive MJ With 0 mg CBD | Inactive MJ With 200 mg CBD | Inactive MJ With 400 mg CBD | Inactive MJ With 800 mg CBD
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 5/50 | 8/50 | 4/50 | 3/50 | 2/50 | 1/50 | 3/50 | 6/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Active MJ With 0 mg CBD (N=50) | Active MJ With 200 mg CBD (N=50) | Active MJ With 400 mg CBD (N=50) | Active MJ With 800 mg CBD (N=50) | Inactive MJ With 0 mg CBD (N=50) | Inactive MJ With 200 mg CBD (N=50) | Inactive MJ With 400 mg CBD (N=50) | Inactive MJ With 800 mg CBD (N=50)
Gastrointestinal Upset (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1/5 (1)
anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold Symptoms (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (foot/hand/tooth) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased heart rate (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No